CLINICAL TRIAL: NCT02143479
Title: A Cohort Study in Liver Transplant Patients Converted From a Tacrolimus Twice a Day (Prograf®) to Tacrolimus Once a Day (Advagraf®). French, Multisite, Observational Study
Brief Title: A Multicenter Study in Liver Transplant Patients Converted From Prograf® to Advagraf® During the First Post-transplantation Year
Acronym: COBALT
Status: Completed | Type: Observational
Sponsor: Astellas Pharma S.A.S. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: FR-ADV-NI-002
Record Dates: First submitted 2014-05-09; First posted 2014-05-21 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2019-03

CONDITIONS: Liver Transplantation
Keywords: France; Prograf; Pharmaco-epidemiology; Tacrolimus; Observational
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1:early conversion from Prograf® to Advagraf®: patients converted from Prograf® to Advagraf® in the first 3 months after transplantation
  Interventions: Drug: Tacrolimus
- 2:late conversion from Prograf® to Advagraf®: patients converted from Prograf® to Advagraf® between 3 months and one year after transplantation
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — oral
  Other Names: FK506; Prograf; Advagraf

SUMMARY:
A study in which two groups of patients will be analysed; patients converted from Prograf to Advagraf within the first 3 months after transplantation and patients converted from Prograf to Advagraf between 3 months and 1 year after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a liver transplant performed in the previous year and for whom the conversion from Prograf® to Advagraf® was decided by the physician.

Exclusion Criteria:

* Patient participating in an interventional clinical trial at the time of enrolment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2014-06-18 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Conversion ratio of the daily dose of tacrolimus (mg Prograf® / mg Advagraf®) | At baseline
  Percentage of patients with a conversion ratio of tacrolimus dose of 1mg/1mg and percentage of patients with a ratio differing from 1mg/1mg
Time of the first tacrolimus trough level (C0) after conversion | From baseline to first determination of C0 (up to 6 months)
  Number of days between the conversion date and the date of the first determination of C0 after conversion
Number of additional visits considered by the physicians to be due to the conversion (if required) | At 6 months and at 1 year follow-up visit
  Percentage of patients with additional visit(s) and percentage of patients without an additional visit

SECONDARY OUTCOMES:
Reasons for conversion | At baseline
  Number of pills, number of treatment intake, treatment compliance, physician request, patient request, safety of treatment, center practice
Patient profile | At baseline
  Sociodemographic data, history of transplantation, comorbidities, complications after transplantation, risk factors, concomitant treatments (other than immunosuppressive protocols) and modification, if required, at 6 months and 1 year after conversion
Collection of immunosuppressive protocol details | At baseline, 6 months and 1 year follow-up visit
  * Date of initiation of treatment with Advagraf®
  * Target tacrolimus C0 (with Prograf® and with Advagraf® and recommendations for administration)
  * Daily dose of Advagraf®
  * Adjustments to Advagraf® dose since the previous visit: date, doses and reason for adjustment
  * Type and dose of immunosuppressive drugs combined with Advagraf®
  * Modification of the immunosuppressive regimen at 6 months and 1 year after conversion (if applicable) since the previous visit: date, modified treatment, type of modification, reason for modification
  * Immunosuppressive regimen at the end of the visit at 6 months and 1 year after conversion, modified treatment, type of modification, reason for modification
Time to reach steady state | From baseline to first determination of C0 (up to 6 months)
Dose ratio at steady state | From baseline and up to 6 months post-conversion
  Ratio of daily dose of tacrolimus during achievement of steady state: mg Prograf® at conversion/mg Advagraf® during achievement of steady state. Percentage of patients with a ratio of 1mg/1mg and percentage of patients with a ratio differing from 1mg/1mg
The Intra -Patient Variability (IPV) of tacrolimus in patients on Prograf® and Advagraf ® | At baseline (Prograf) and during the 45 days after conversion (Advagraf)
Latest available laboratory data with Prograf® before conversion and with Advagraf® | At baseline, 6 months and 1 year follow-up visit
  Values and dates for renal parameters, liver parameters, blood glucose and Hepatitis C viral load
Compliance with treatment at conversion | At baseline and at 1 year after conversion
  Compliance with treatment at conversion (with Prograf® and only in group 2) and at 1 year after conversion (with Advagraf® for both groups) will be assessed using the Morisky questionnaire and a score will be calculated
Patients' quality of life at conversion | At baseline and at 1 year after conversion
  Patients' quality of life at conversion (with Prograf® only in group 2) and at 1 year after conversion (with Advagraf® for both groups) will be assessed using the European Quality of Life-5 Dimensions 5 level (EQ5D-5L) questionnaire
Rate of acute rejection proven by biopsy (BPAR), graft survival rate and patient survival rate | 6 months and 1 year
  Will be assessed on the basis of the number of acute rejections confirmed by biopsy and recorded adverse events and adverse reactions
Occurrence of adverse events and/or effects | From baseline until 1 year follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical and Scientific Affairs Manager, Transplantation, Study Director — Astellas Pharma S.A.S.
Locations (17):
- France (17):
  - Site, Besançon
  - Site, Bordeaux
  - Site, Caen
  - Site, Chambray-lès-Tours
  - Site, Clichy
  - Site, Créteil
  - Site, Grenoble
  - Site, Lille
  - Site, Limoges
  - Site, Lyon
  - Site, Marseille
  - Site, Montpellier
  - Site, Nice
  - Site, Paris
  - Site, Rennes
  - Site, Toulouse
  - Site, Villejuif

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.